CLINICAL TRIAL: NCT03782467
Title: A First-in-human, Multicenter, Open-label, Phase 1 Study in Patients With Advanced and/or Refractory Solid Malignancies to Evaluate the Safety of Intravenously Administered ATOR-1015
Brief Title: Phase 1 Study in Patients With Advanced and/or Refractory Solid Malignancies to Evaluate the Safety of ATOR-1015
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-18-1015-C-01
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumor; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATOR-1015 (Experimental): ATOR-1015 administered by intravenous infusions every 2 weeks until confirmed progressive disease, unacceptable toxicity or withdrawal of consent.
  Interventions: Biological: ATOR-1015

INTERVENTIONS:
Biological: ATOR-1015 — Bispecific human monoclonal antibody targeting cytotoxic T-lymphocyte associated protein 4 (CTLA-4) and OX40 (also known as CD134)

SUMMARY:
The aim of the study is to investigate the safety and tolerability of ATOR-1015 when administered as repeated intravenous infusions to patients with advanced and/or refractory solid malignancies.

ELIGIBILITY:
Major Inclusion Criteria:

* Diagnosis of advanced and/or refractory solid malignancy
* Eastern Cooperation Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months

Major Exclusion Criteria:

* Organ transplant recipient
* Active autoimmune disorder
* Other malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AEs) assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | From start of study until 28 days after last dose
  Number of participants with treatment-related AEs assessed by CTCAE v5.0
Safety and tolerability: Vital signs | From start of study until end of study (28-56 days after last dose)
  Vital signs include blood pressure, pulse rate, oxygen saturation and body temperature. Clinically significant abnormal findings will be reported as AEs.
Safety and tolerability: Physical examination | From start of study until end of study (28-56 days after last dose)
  Physical examination will as a minimum include examination of mouth, throat, lymph nodes, respiratory, cardiovascular system, abdomen, extremities, neurological system and skin. Clinically significant abnormal findings will be reported as AEs.
Safety and tolerability: 12-lead electrocardiogram (ECG) | From start of study until end of study (28-56 days after last dose)
  Clinically significant abnormal ECG findings will be reported as AEs.
Safety and tolerability: Clinical laboratory tests | From start of study until end of study (28-56 days after last dose)
  Clinical laboratory tests include clinical chemistry, hematology, coagulation, hormones and urinalysis.

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum observed serum concentration of ATOR-1015 (Cmax) | From start of study until end of study (28-56 days after last dose)
Pharmacokinetics: Time to Cmax | From start of study until end of study (28-56 days after last dose)
Pharmacokinetics: Area under the ATOR-1015 serum concentration-time curve (AUC) | From start of study until end of study (28-56 days after last dose)
Immunogenicity: Anti-drug antibody (ADA) titer in serum | From start of study until end of study (28-56 days after last dose)
  Levels of antibodies to ATOR-1015 will be evaluated
Clinical efficacy: Anti-tumor activity assessed by response evaluation criteria in solid tumors for immune-based therapeutics (iRECIST) | From start of study until end of study (28-56 days after last dose)
  Computed tomography (CT) scans of tumors will be evaluated according to iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Malin Carlsson, MD, Study Director — Alligator Bioscience AB; Jeffrey Yachnin, Dr, Principal Investigator — Centrum för Kliniska Cancerstudier (CKC), Karolinska Universitetssjukhuset
Locations (5):
- Denmark (2):
  - Phase 1 Unit, Department of Oncology, Rigshospitalet, Copenhagen
  - Center for Cancer Research, Department of Oncology, Herlev Hospital, Herlev
- Sweden (3):
  - Kliniska Prövningsenheten, Kliniska Studier Sverige - Forum Söder, Skånes Universitetssjukhus, Lund
  - Centrum för Kliniska Cancerstudier (CKC), Fas 1-enheten, Karolinska Universitetssjukhuset, Solna
  - Onkologavdelningen, Akademiska Sjukhuset, Uppsala

REFERENCES:
- [Derived] Kvarnhammar AM, Veitonmaki N, Hagerbrand K, Dahlman A, Smith KE, Fritzell S, von Schantz L, Thagesson M, Werchau D, Smedenfors K, Johansson M, Rosen A, Aberg I, Winnerstam M, Nyblom E, Barchan K, Furebring C, Norlen P, Ellmark P. The CTLA-4 x OX40 bispecific antibody ATOR-1015 induces anti-tumor effects through tumor-directed immune activation. J Immunother Cancer. 2019 Apr 11;7(1):103. doi: 10.1186/s40425-019-0570-8. PMID 30975201